CLINICAL TRIAL: NCT01142154
Title: A Phase I/II Crossover Study To Evaluate and Compare the Pharmacokinetics of a Single IV Dose of D-Mannitol (Osmitrol®10%) to Single and Multiple, Escalating Doses of Liquid, Oral Prodarsan™ in Patients With Cockayne Syndrome
Brief Title: Pharmacokinetics and Safety Study of Single and Multiple Oral Doses Prodarsan™ in Patients With Cockayne Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: DNage B.V. (Industry)
Responsible Party: Lia Dam/Director Clinical Operations, DNage
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MP1104-02
Record Dates: First submitted 2010-05-20; First posted 2010-06-11 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Cockayne Syndrome
Keywords: Cockayne Syndrome; Ageing; pediatrics; Pharmacokinetics; Prodarsan; Dwarfism; Genetic disease, inborn; DNA Repair-Deficiency Disorders; Tolerability; Safety
MeSH Terms: conditions — Cockayne Syndrome; Dwarfism; Genetic Diseases, Inborn; DNA Repair-Deficiency Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- oral, liquid solution (Experimental)
  Interventions: Drug: Prodarsan

INTERVENTIONS:
Drug: Prodarsan — Prodarsan TID, oral solution, 6-8 days

SUMMARY:
This study is to compare the exposure of orally administered Prodarsan to the intravenous dosed Osmitrol (10% solution) in Cockayne Syndrome (CS) patients. Also the pharmacokinetics of single and multiple orally dosed Prodarsan will be evaluated and compared to intravenous dose of Osmitrol in CS patients.

ELIGIBILITY:
Inclusion Criteria:

* Parents or legal guardian(s) of the pediatric patient with CS must be willing and able to give written Informed Consent. Informed Assent will be offered to children who can understand and participate in the Informed Assent process.
* Diagnosis of CS confirmed by one of the following laboratory diagnostic test results:

  * Demonstration by molecular diagnostic analyses of two mutations in either the ERCC6 gene or the ERCC8 gene, wherein both mutations are either known to be pathogenic or are obviously detrimental (including nonsense or frameshift mutations, mutations of "invariant" splice site consensus signals, or large deletions/rearrangements); OR
  * A pattern of DNA repair responses in patient's cultured skin fibroblast cells indicative of a specific deficiency of transcription-coupled DNA nucleotide excision repair after irradiation with ultraviolet light, namely a significant deficiency of cellular survival (and/or "recovery of ribonucleic acid [RNA] synthesis," if that has been specifically measured) coupled with a normal test for "unscheduled DNA synthesis" OR
  * Decreased cell survival and/or "recovery of RNA synthesis" in UV-irradiated patient's skin fibroblast cultures and rescue of these parameters by fusion to reference cell lines with known NER defects (functional complementation analysis) OR
  * Quantitative RT-PCR to quantify mRNA levels of CS-A and CS-B transcripts.
* Weight inclusive of 10 kg to 25 kg.
* Male or female, inclusive of two (2) to ten (10) years of age.
* Clinically acceptable hematocrit as judged by the Principal Investigator (PI).
* The investigator has the opinion that the patient and caregiver are willing and able to comply with protocol requirements.

Exclusion Criteria:

* Any concurrent illness (other than related to CS), disability or clinically significant abnormality, including laboratory tests, that may affect the interpretation of the PK or safety data or prevent the patient from safely completing the assessments required by the protocol as judged by the investigator. Such conditions include, but are not limited to:

  * Ascites or generalized edema.
  * Nephrotic syndrome or history of abnormal kidney function.
  * Clinically significant thyrotoxicosis.
  * Known history of hyperprolinemia.
  * Clinically significant dehydration as judged by the investigator
* Severely compromised venous access.
* Presence of an external ventricular, abdominal, or chest drain.
* Subjects due to receive radioiodine therapy, two (2) weeks before or two (2) weeks following the study period.
* Participation in another PK or treatment clinical study within thirty (30) days prior to signing and dating of Informed Consent/Assent Form for this study.
* As judged by the investigator, clinical features present at the time of initial screening, that are associated with the terminal phases of the natural progression of CS, indicating that safe travel and completion of the study and its assessments are unlikely, including any of the following:

  * Continuous or intermittent dependence on supplemental oxygen at home during the six (6) months prior to enrollment in this study; OR
  * Two or more hospitalizations due to pneumonia, during the twelve (12) months prior to enrollment in this study; OR
  * A documented, net weight loss of at least 10%, which has not been recovered, and which includes a significant net weight loss (beyond the estimated error of the measurement) over the most recent 6 months despite intensive nutritional support including the use of gastrostomy tube feedings.
* Known hypersensitivity to any of the components found in Prodarsan, D-mannitol, iohexol or iodine compounds.
* History of clinically significant drug sensitivity or allergic reaction such as anaphylaxis.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Evaluate and compare the pharmacokinetics of D-mannitol following a single IV dose of Osmitrol to single and multiple oral doses of Prodarsan in pediatric patients with Cockayne Syndrome | 6 months

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of administering oral Prodarsan in CS patients over a six (6) to eight (8) day period, including dose escalation to reach a Target Dose | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Edward Neilan, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States